CLINICAL TRIAL: NCT04712448
Title: Serum Prevalence of Antibodies Anti-SARS-Cov-2 in Healthy Subjects and in Patients With Chronic Diseases in Pre-pandemic Blood Samples
Brief Title: Serum Prevalence of SARS-Cov-2 Antibodies in Pre-pandemic Blood Samples (SPARE)
Acronym: SPARE
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Department of Transfusion Medicine Venice Area (Unknown); Istituto per lo Studio, la Prevenzione e la Rete Oncologica (Other)
Responsible Party: Sponsor
Other Study IDs: 20/33
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Healthy; Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum and whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Donors of the Transfusion Center of Venice Healthy volunteers afferent to BioBIM
  Interventions: Diagnostic Test: Anti-COVID test
- Patients: Patients with chronic diseases afferent to BioBIM
  Interventions: Diagnostic Test: Anti-COVID test

INTERVENTIONS:
Diagnostic Test: Anti-COVID test — No intervention is foreseen by the protocol

SUMMARY:
The first reports of infections caused by SARS-CoV-2 were released from Wuhan, China in December 2019. From there, the infection quickly spread into a pandemic form. The clinical manifestation of the infection varies enormously, from totally asymptomatic or mildly symptomatic forms, with nonspecific and flu-like manifestations, to an acute respiratory distress syndrome which, in patients requiring hospitalization in the ICU and mechanical ventilation invasive, can lead to death, especially in elderly subjects and carriers of co-morbidities. Recently, the association of blood groups ABO as possible biological markers of susceptibility to COVID-19, has been evaluated, linking blood type O with a lower chance of infection, blood type A with the highest risk, and blood group B with the greatest complications.

In Italy, the first non "imported" case dates back to February 2020, although new evidence on subjects tested positive for the antibody assay on serum samples suggests that the virus started to circulate before the official date.

Few are the data relating to asymptomatic infections or with mild non-specific and nuanced symptoms that have been quantified in about 85% of the total number of infected. Moreover, thanks to the availability of serological tests that identify the presence of anti-SARS-CoV-2 antibodies, it emerged that a proportion of the population was infected by the virus and developed an antibody response and that almost 30% of the people with antibodies were asymptomatic. In order to evaluate the seroprevalence of COVID-19 infection among asymptomatic subjects the investigators will conduct specific serological tests (total antibodies) to identify the prevalence of SARS-2-CoV antibodies among healthy blood donors who went to transfusion facilities of the DIMT in Venice during the pandemic (about 2500 periodic donors who referred to the Transfusion Center in the period between May and October 2019). Patients afferent to the Interinstitutional Multidisciplinary Biobank (BioBIM) of the Research Center of the IRCCS San Raffaele Pisana in Rome, with or without concomitant co-morbidities (about 1000 subject) will be also tested. All samples will be analyzed for any association with sex, age group and blood group.

DETAILED DESCRIPTION:
1. Title Serum prevalence of SARS-Cov-2 antibodies in pre-pandemic blood samples
2. Background The first reports of infections caused by SARS-CoV-2, a Beta Corona virus, single-stranded RNA, were released from Wuhan, China in December 2019. From there, the infection quickly spread into a pandemic form.

   The clinical manifestation of the infection varies enormously, from totally asymptomatic or mildly symptomatic forms, with nonspecific and flu-like manifestations, to an acute respiratory distress syndrome which, in patients requiring hospitalization in the ICU and mechanical ventilation invasive, can lead to death. The greater severity of the course of the infection depends greatly on the general conditions of the patients, being maximum in elderly subjects and carriers of co-morbidities. Recent studies have also evaluated the association of blood groups ABO as possible biological markers of susceptibility to COVID-19, suggesting that people with blood type O have a lower chance of infection while individuals with blood type A are most at risk, and people with blood group B have the greatest complications in the event of infection.

   In Italy, the first non "imported" case dates back to February 2020 in a person residing in Lombardy, in the province of Lodi. However, new evidence on subjects tested positive for the antibody assay on serum samples suggests that the virus started to circulate before the official date.

   Initially, due to the sudden explosion of cases, epidemiological surveillance focused on patients related to health facilities because they were symptomatic, suspicious and high-risk contacts. Few are the data relating to asymptomatic infections or with mild non-specific and nuanced symptoms that, data from China, would quantify in about 85% of the total number of infected. Precisely on the role of person-to-person transmission in the course of asymptomatic infection and in the subclinical phases of the disease, epidemiological data are lacking despite they could prove to be very important. In fact, thanks to the availability of serological tests that identify the presence of anti-SARS-CoV-2 antibodies, it emerged that a proportion of the population was infected by the virus and developed an antibody response and that almost 30% of the people with antibodies were asymptomatic. Therefore, the understanding of the prevalence of the disease and the prevalence of the antibody response appear to be of considerable interest, as it seems to be established that asymptomatic subjects can transmit the SARS-CoV-2 infection for a period that in some cases has proved greater than 14 days.

   In order to evaluate the seroprevalence of COVID-19 infection among asymptomatic subjects, thus obtaining a real estimate of the beginning of the circulation of the virus in Italy, in the present study the investigators intend to conduct specific serological tests (total antibodies) to identify the prevalence of SARS-2-CoV antibodies among healthy blood donors who went to transfusion facilities of the DIMT in Venice during the pandemic (about 2500 periodic donors who referred to the Transfusion Center in the period between May and October 2019).

   Samples belonging to healthy volunteers (about 500) who have agreed to donate their blood will also be evaluated to establish a pool of control subjects belonging to the Interinstitutional Multidisciplinary Biobank (BioBIM) of the Research Center of the IRCCS San Raffaele Pisana in Rome. Finally, in order to evaluate the impact of seroprevalence in subjects with chronic diseases (about 1000), such as cardiovascular, oncological, respiratory and neurodegenerative ones, which represent settings of COVID-19 positive patients with a poorer prognosis, patient samples with the listed comorbidities, already present in BioBIM, will be analyzed. It has recently emerged that seroprevalence increases with increasing age and that younger groups have a lower susceptibility to infection. Therefore, all samples will be analyzed for any association with sex, age group and blood group.
3. Promoter Prof.ssa Fiorella Guadagni
4. Sponsor/Promotor IRCCS San Raffaele Pisana
5. Site IRCCS San Raffaele Pisana
6. Study type Multicentric, retrospective, observational, non pharmacological, on biological samples, conducted at the IRCCS San Raffaele Pisana, Rome, aimed at verifying the seroprevalence of SARS-COV-2 antibodies in the population.
7. Objectives 7.1 PRIMARY Objective: The aim of the study is to determine the proportion of people in the general population who developed an antibody response to antigenic determinants of SARS-CoV-2 in the period preceding the spread of the virus in Italy.

   7.2 SECONDARY Objective: Secondary objectives are represented by the possibility to characterize the differences in prevalence between genders, age groups and blood groups, also in relation to more unfavourable courses in subjects with other chronic diseases.
8. Participants

   The study protocol will involve a total of 3500 subjects (3000 healthy subjects and 1000 patients with chronic diseases) aged> 18 years, of both sexes. The two groups will be formed as follows:

   A- Healthy subjects among periodic blood donors of the Transfusion Center and volunteer donors of BioBIM B- Patients with chronic diseases including cardiovascular, respiratory, oncological and neurodegenerative diseases related to BioBIM
9. Inclusion/exclusion Criteria 9.1 Inclusion criteria - Both sexes

   * Age >18 years
   * Signed informed consent for the donation / sample storage in the Biological Bank 9.2 Exclusion criteria
   * for healthy subjects, all those who have shown any symptoms, albeit mild, in the 28 days prior to the donation.
   * patients who have not signed the informed consent for the conservation of their samples in the Biological Bank.

   9.3 Drop out Not applicable.
10. Study design

    The study will last 9 months, and includes 3 phases as follows:

    Phase 1: identification of samples Phase 2: sample analysis Phase 3: statistical analysis
11. Methods of contact with possible participants in the study Not applicable. The study will be carried out only on samples stored in the Biobank.
12. Methods of acquisition, statistical analysis of data and storage of raw data, compliance with privacy regulations Data collection will be carried out on a dedicated and anonymized database by the Principal Investigator. Data will be stored on a dedicated and protected server.
13. Statistical Methodology 13.1 Statistical analysis Statistical analysis of all parameters will be conducted under the responsibility of the Biomarker Discovery and Advanced Technologies (BioDAT) Unit of IRCCS San Raffaele Pisana.

Data analysis will be carried out using frequency and percentage for the categorical variables, and mean and standard deviation for the quantitative variables. The t-test will be used to compare means and a p-value less than 0.05 will be considered statistically significant. All analysis will be performed on the SPSS Statistical Package for Social Sciences.

13.2 Sample size The SPARE study is a pilot study, designed to verify the adequacy and feasibility of the project, and to obtain preliminary data that allow to determine the size of the sample of the final study. The sample size is therefore represented by a consecutive number of subjects who donated blood in the period May-October 2019 (about 2500) and all subjects (healthy and with chronic diseases) who referred to BioBIM in 2019 (about 1500 ).

14) Requirements of originality and scientific soundness of the study The SPARE study aims to evaluate the seroprevalence of COVID-19 infection among asymptomatic subjects and thus obtain a real estimate of the beginning of the circulation of the virus in Italy. The evidence currently present in the literature refers mainly to the period of the actual pandemic, but there are no data relating to the months prior to autumn 2019. Same for the official data released by the Ministry of Health in collaboration with the National Institute of Statistics (ISTAT). This study will allow us to define the spread of the SARS-2-CoV virus in a period long before the date to which the pandemic began in Italy.

15) Expected Results

The main expected results are:

1. Identification of seroprevalence of anti-SARS-2-CoV antibodies in the population prior to the date on which the beginning of the infection in Italy is officially traced;
2. Description of any associations with sex, age, blood group, outcomes of patients with chronic diseases.

16) Progress report The proposers will submit a report on the progress of the study to the Ethics Committee at the end of each year and at the end of the study.

17) Feasibility

- n. patient samples that may be included is consistent with the study design

* presence of the necessary equipment
* adequacy of personnel 18) Concomitant treatments Not applicable. The SPARE study is a study on biological samples only 19) Cost/benefit ratio The study is supported by the IRCCS San Raffaele Pisana. The inclusion of samples belonging to healthy donors and patients in this clinical study may provide benefits in terms of more accurate management and acquisition of indications on the spread of the Sars-COV-2 virus in the asymptomatic population. There are no risks.

  20) Ethical relevance The study is conducted on patient samples stored in the Biological Banks, therefore there are no problems of an ethical nature to its execution.

  21) Insurance The procedures provided for the study in this centre do not directly involve patients, but the analysis of samples taken in the centres they enrol. The researcher assigned to the analysis of the samples is covered by an insurance policy included in the contract stipulated with the IRCCS San Raffaele Pisana.

  22) Result publication In compliance with the provisions in force regarding the confidentiality of sensitive data and patent protection, the results of the study will be submitted for publication within 6 months of after the closure of the database.

  23) Informed Consent The submission of specific informed consent for this study on anonymized samples from biological banks or large collections does not apply.

  24) Ethical aspects This protocol will be conducted in accordance with the ethical principles that draw their origin from the Declaration of Helsinki, respects the GCP and applicable regulatory provisions.

  25) References
  1. Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, et al. China Novel Coronavirus Investigating and Research Team A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020;382(8):727-33. 10.1056/NEJMoa2001017
  2. World Health Organization (WHO). Novel coronavirus - China. Geneva: WHO; 12 Jan 2020. [Accessed 09 Oct 2020]. Available from: https://www.who.int/csr/don/12-january-2020-novel-coronavirus-china/en/
  3. Santos-Sánchez NF, Salas-Coronado R. Medwave. Origin, structural characteristics, prevention measures, diagnosis and potential drugs to prevent and COVID-19. 2020 Sep 25;20(8):e8037. doi: 10.5867/medwave.2020.08.8037.
  4. Luo L, Fu M, Li Y, Hu S, Luo J, Chen Z, Yu J, Li W, Dong R, Yang Y, Tu L, Xu X. The potential association between common comorbidities and severity and mortality of coronavirus disease 2019: A pooled analysis. Clin Cardiol. 2020 Oct 7. doi: 10.1002/clc.23465.
  5. Zaho J, Yang Y, Huang H, Li D, Gu D., Lu X, et al. Relationship between the ABO Blood Group and the COVID-19 susceptibility. 10.1101/2020.03.11.20031096
  6. Zalba Marcos S, Luisa Antelo M, Galbete A, Etayo M, Ongay E, García-Erce JA. Infection and thrombosis associated with COVID-19: Possible role of the ABO blood group. Med Clin (Engl Ed). 2020 Sep 26. doi: 10.1016/j.medcle.2020.06.013.
  7. Livingston E, Bucher K. Coronavirus Disease 2019 (COVID-19) in Italy. JAMA. 2020;323(14):1335. 10.1001/jama.2020.4344
  8. Mizumoto K, Kagaya K, Zarebski A, Chowell G. Estimating the asymptomatic proportion of coronavirus disease 2019 (COVID-19) cases on board the Diamond Princess cruise ship, Yokohama, Japan, 2020. Euro Surveill 2020;25(10):2000180.
  9. ISTAT. Primi risultati dell'indagine di sieroprevalenza sul SARS-CoV-2. Accessible presso https://www.istat.it/it/archivio/246156
  10. Oran DP, et al. Prevalence of Asymptomatic SARS-CoV-2 Infection - A Narrative Review. Ann Int Med 2020; 173:362-376. doi.org/10.7326/M20-3012.
  11. Pagani G, et al. Seroprevalence of SARS-CoV-2 significantly varies with age: Preliminary results from a mass population screening. J Infect. 2020 Sep 19;S0163-4453(20)30629-0. doi: 10.1016/j.jinf.2020.09.021.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age >18 years
* Signed informed consent for the donation / sample storage in the Biological Bank

Exclusion Criteria:

* for healthy subjects: all those who have shown any symptoms, albeit mild, in the 28 days prior to the donation.
* for patients: who have not signed the informed consent for the conservation of their samples in the Biological Bank.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study protocol will involve a total of 3500 subjects (3000 healthy subjects and 1000 patients with chronic diseases) aged> 18 years, of both sexes. The two groups will be formed as follows:
  A- Healthy subjects among periodic blood donors of the Transfusion Center and volunteer donors of BioBIM B- Patients with chronic diseases including cardiovascular, respiratory, oncological and neurodegenerative diseases related to BioBIM
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence of antibodies anti-COVID-19 | May-October 2019
  Seroprevalence of antibodies anti-COVID-19

SECONDARY OUTCOMES:
Correlation with blood group | May-October 2019
  Correlation with blood group

OTHER OUTCOMES:
Correlation with co-morbidities | May-October 2019
  Correlation with co-morbidities

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Rome, Italy